CLINICAL TRIAL: NCT02285634
Title: The Effect of Intranasal Vasoconstrictor Medications on Hemodynamic Parameters: A Randomized Double-blind, Placebo-controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias Kummer, Assistant Professor of Emergency Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-006312; UL1TR000135 (NIH)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Epistaxis; Blood Pressure
MeSH Terms: conditions — Epistaxis | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxymetazoline 0.05% (Experimental): Oxymetazoline 0.05%
  Interventions: Drug: Oxymetazoline 0.05%
- Phenylephrine 0.25% (Experimental): Phenylephrine 0.25%
  Interventions: Drug: Phenylephrine 0.25%
- Lidocaine 1% plus epinephrine 1:100,000 (Experimental): Lidocaine 1% plus epinephrine 1:100,000
  Interventions: Drug: Lidocaine 1% plus epinephrine 1:100,000
- Bacteriostatic 0.9% sodium chloride (NaCL) (Placebo Comparator): Bacteriostatic 0.9% NaCL
  Interventions: Drug: Bacteriostatic 0.9% NaCL

INTERVENTIONS:
Drug: Oxymetazoline 0.05% — sterile gauze soaked in 5 milliliters (mL) of Oxymetazoline 0.05% into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
  Arms: Oxymetazoline 0.05%
Drug: Phenylephrine 0.25% — sterile gauze soaked in 5 milliliters (mL) of Phenylephrine 0.25% into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
  Arms: Phenylephrine 0.25%
Drug: Lidocaine 1% plus epinephrine 1:100,000 — sterile gauze soaked in 5 milliliters (mL) of Lidocaine 1% plus epinephrine 1:100,000 into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
  Arms: Lidocaine 1% plus epinephrine 1:100,000
Drug: Bacteriostatic 0.9% NaCL — sterile gauze soaked in 5 milliliters (mL) of Bacteriostatic 0.9% NaCL into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
  Arms: Bacteriostatic 0.9% sodium chloride (NaCL)

SUMMARY:
Nosebleeds (epistaxis) are a frequent cause of emergency department visits, reportedly inciting 1 in 200 visits. They are most common in those less than ten and older than seventy, often occurring in the winter months secondary to dry indoor heating. Epistaxis is associated with elevated blood pressures, but it is controversial whether hypertension is actual a contributing cause.

In non-life-threatening epistaxis, the first step in management is commonly the application of a topical vasoconstrictive medication. In many cases this will lead to cessation of the bleeding or facilitate the exam in those that continue to bleed. Frequently used medications include phenylephrine, oxymetazoline, and lidocaine with epinephrine.

Classic teaching has been to avoid the use of these medications in patients with elevated blood pressures due to concerns of inducing hypertensive crisis. Strict avoidance of topical vasoconstrictors in this patient group with epistaxis severely limits the treatment options for a many patients given the association between the two conditions.

Though universally taught, the actual effect of these agents on blood pressure remains unquantified. Studies investigating the prevention of nose bleeding during nasotracheal intubations suggest that the effect might be minor with little variation between agents.

Clinical question:

What is the effect of commonly used intranasal vasoconstrictors on blood pressure in volunteers without a history of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over the age of eighteen that have been recently dismissed from the Emergency Department at Mayo Clinic Hospital, Saint Marys Campus.
* We will recruit a convenience sample of 100 patients from the Emergency Department who have completed their Emergency Department evaluation and treatment and are being discharged to home with non-painful conditions.

Exclusion Criteria:

* We will exclude persons under the age of eighteen
* Vulnerable populations (pregnant patients and prisoners)
* Those with an allergy to any of the study agents
* Those with acute pain
* Those using antihypertensive or antiarrhythmic agents
* Those with significant cardiopulmonary comorbidities (namely history of arrhythmia, coronary artery disease, hypertension, and heart failure)
* Those with concomitant use of Monoamine oxidase A (MAO) Inhibitors
* Those with a diagnosis of angle closure glaucoma or benign prostatic hyperplasia (BPH)
* Those with a history of cerebrovascular disease
* As well as those with a history of previous nasal surgery or known nasal anatomic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kummer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellew SD, Johnson KL, Nichols MD, Kummer T. Effect of Intranasal Vasoconstrictors on Blood Pressure: A Randomized, Double-Blind, Placebo-Controlled Trial. J Emerg Med. 2018 Oct;55(4):455-464. doi: 10.1016/j.jemermed.2018.07.004. Epub 2018 Sep 6. PMID 30195946
- See also: The Journal of Emergency Medicine — https://doi.org/10.1016/j.jemermed.2018.07.004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers over the age of eighteen that have been recently dismissed from the Emergency Department at Mayo Clinic Hospital, Saint Marys Campus beginning 11-12-14.
Pre-assignment Details: None to report
Groups:
- Bacteriostatic 0.9% Sodium Chloride (NaCL): Bacteriostatic 0.9% NaCL
  Bacteriostatic 0.9% sodium chloride (NaCL): sterile gauze soaked in 5 milliliters (mL) of Bacteriostatic 0.9% NaCL into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
Period: Overall Study
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% Sodium Chloride (NaCL)
Started | 15 | 20 | 15 | 18
Completed | 15 | 20 | 11 | 17
Not Completed | 0 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bacteriostatic 0.9% NaCL: Bacteriostatic 0.9% sodium chloride (NaCL)
  Bacteriostatic 0.9% sodium chloride (NaCL): sterile gauze soaked in 5 milliliters (mL) of Bacteriostatic 0.9% NaCL into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
- Total: Total of all reporting groups
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL | Total
Number analyzed (Participants) | 15 | 20 | 11 | 17 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (15.0) | 40.0 (16.8) | 38.6 (15.7) | 31.2 (10.1) | 36.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 2 | 8 | 29
  Male | 4 | 12 | 9 | 9 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 20 | 11 | 17 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Blood Pressure
Description: Change in mean arterial blood pressure from the baseline measurement
Time Frame: baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL
Number analyzed (Participants) | 15 | 20 | 11 | 17
mmHg | 5.1 (6.8) | 6.4 (5.8) | 4.6 (8.0) | 6.5 (5.5)
Statistical Analysis 1: Comparison: Lidocaine 1% Plus Epinephrine 1:100,000 vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.42, Fisher Exact
Statistical Analysis 2: Comparison: Oxymetazoline 0.05% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.52, Fisher Exact
Statistical Analysis 3: Comparison: Phenylephrine 0.25% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.93, Fisher Exact

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change from baseline in systolic blood pressure.
Time Frame: baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Bacteriostatic 0.9% NaCL: Bacteriostatic 0.9% sodium chloride (NaCL)
  Bacteriostatic 0.9% NaCL: sterile gauze soaked in 5 milliliters (mL) of Bacteriostatic 0.9% sodium chloride (NaCL) into one nostril and placement of a nasal clamp. The nasal clamp and medication will be removed after 15 minutes.
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL
Number analyzed (Participants) | 15 | 20 | 11 | 17
mmHg | 7.5 (9.8) | 8.2 (7.2) | 3.5 (6.5) | 8.9 (5.4)
Statistical Analysis 1: Comparison: Lidocaine 1% Plus Epinephrine 1:100,000 vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.06, Fisher Exact
Statistical Analysis 2: Comparison: Oxymetazoline 0.05% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.61, Fisher Exact
Statistical Analysis 3: Comparison: Phenylephrine 0.25% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.78, Fisher Exact

3. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change from baseline in diastolic blood pressure.
Time Frame: baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL
Number analyzed (Participants) | 15 | 20 | 11 | 17
mmHg | 5.7 (7.7) | 7.9 (6.8) | 6.2 (8.3) | 9.3 (6.6)
Statistical Analysis 1: Comparison: Lidocaine 1% Plus Epinephrine 1:100,000 vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.27, Fisher Exact
Statistical Analysis 2: Comparison: Oxymetazoline 0.05% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.17, Fisher Exact
Statistical Analysis 3: Comparison: Phenylephrine 0.25% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.56, Fisher Exact

4. Secondary Outcome: Change in Heart Rate
Description: Change from baseline in heart rate.
Time Frame: baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL
Number analyzed (Participants) | 15 | 20 | 11 | 17
beats/min | 2.8 (5.2) | 5.2 (6.6) | 7.5 (9.7) | 6.8 (5.6)
Statistical Analysis 1: Comparison: Lidocaine 1% Plus Epinephrine 1:100,000 vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.78, Fisher Exact
Statistical Analysis 2: Comparison: Oxymetazoline 0.05% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.10, Fisher Exact
Statistical Analysis 3: Comparison: Phenylephrine 0.25% vs Bacteriostatic 0.9% NaCL; Test type: Superiority; p = 0.47, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study protocol. Total observation time was 30 minutes and after completion of the study protocol any adverse effects were recorded.
Arm/Group | Oxymetazoline 0.05% | Phenylephrine 0.25% | Lidocaine 1% Plus Epinephrine 1:100,000 | Bacteriostatic 0.9% NaCL
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/20 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 4/15 | 3/20 | 0/11 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxymetazoline 0.05% (N=15) | Phenylephrine 0.25% (N=20) | Lidocaine 1% Plus Epinephrine 1:100,000 (N=11) | Bacteriostatic 0.9% NaCL (N=17)
Nasal Pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Eye watering (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unpleasant aftertaste (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The primary limitation was the small sample size as enrollment was markedly more difficult than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes